CLINICAL TRIAL: NCT07382739
Title: A Phase 2 Study of Radiotherapy-induced Immune Priming to Enhance Elranatamab (Elra) in Relapsed Refractory Multiple Myeloma (RRMM) With Extramedullary Disease (EMD) and Paramedullary Disease (PMD) "PRIME-EMD-PMD"
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1557; NCI-2026-00668 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Phase 2; Radiotherapy-Induced Immune Priming; Elranatamab; Relapsed Refractory Multiple Myeloma (RRMM); Extramedullary Disease in Multiple Myeloma; Paramedullary Disease; PMD
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with Elranatamab (SubQ) Q4W (Experimental): To evaluate the efficacy of RT-induced immune priming to enhance Elranatamab (Elra) in RRMM with EMD or PMD as measured by overall response rate
  Interventions: Drug: Elranatamab

INTERVENTIONS:
Drug: Elranatamab — Given by IV

SUMMARY:
To learn if low doses of radiation therapy can help the drug elranatamab enhance the killing effect of the cancer cells.

DETAILED DESCRIPTION:
Primary Objectives To evaluate the efficacy of RT-induced immune priming to enhance Elranatamab (Elra) in RRMM with EMD or PMD as measured by overall response rate (ORR) at 3 months

Secondary Objectives To describe adverse events (AEs). To determine time to next treatment (TTNT). To evaluate progression-free survival (PFS). To determine overall survival (OS). To estimate quality of life (QOL). To assess local control to the irradiated lesions To determine differences in response in patients with EMD vs PMD To determine differences in response in patients High Risk (HR) vs Standard Risk (SR) disease

ELIGIBILITY:
Inclusion Criteria

* RRMM exposed to IMID, PI, anti-CD38 mAb, relapsed or refractory to at least one prior line of therapy (LOT), progressed on or after the last regimen:

  1. Relapsed disease: progressive disease (PD) >60 days after cessation of prior therapy
  2. Refractory disease: PD <=60 days after cessation of prior therapy, <25% reduction in paraprotein (monoclonal protein [M-protein] or serum free light chains [sFLC]) or measurements of EMD/PMD
* Diagnosis of relapsed or refractory multiple myeloma as indicated by progression by IMWG criteria
* At least one locus of EMD or PMD present on imaging (either PET/CT or magnetic resonance imaging [MRI]):
* EMD: extramedullary plasmacytoma, not a contiguous extension from a bone lesion.
* PMD: paraskeletal plasmacytoma, contiguous extension from a bone lesion At least one locus of EMD/PMD that was not previously radiated and can be treated with radiation
* Hematology (supportive care is allowed, including transfusions and granulocyte colony stimulating factor (G-CSF), if cytopenia is deemed secondary to myeloma disease burden):
* Hemoglobin (Hgb) >=7g/dL
* Platelet>=50K/uL
* Absolute neutrophil count (ANC) >=0.75K/uL
* Chemistry:
* Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) <=2.5 x upper
* limit of normal (ULN)
* Total bilirubin (TBili) <=1.5ULN (except for a known history of Gilbert syndrome)
* Creatinine clearance (CrCL) >=30mL/min/1.73m2
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) <=2, unless ECOG PS due to pain/morbidity secondary to underlying myeloma disease, with the potential of improved ECOG PS to <=2.
* All participants must be either
* Not of childbearing potential, or
* Practicing at least 1 highly effective method of contraception until 6 months after the last dose of study treatment.
* Childbearing age female participantsmust have a negative serum pregnancy test at screening and must agree to further pregnancy tests during the study.

Exclusion Criteria

1. Prior or concurrent exposure to any of the following in the specified time frame prior to the first dose of Elra treatment:

   * Within 14 days or at least 5 half-lives, whichever is less, of any investigational treatment
   * Within 7 days of IMIDs, PI, anti-CD38 mAb, or cytotoxic systemic myeloma therapies
   * Within 12 weeks of autologous stem-cell therapy (ASCT) or 6 months of AlloSCT and has to be off immunosuppressive agents >=42 days without signs of graft versus host disease (GVHD)
   * Within 2 weeks of major surgery
   * Within 6 months of cerebrovascular accident (CVA) events
2. Waldenstrom, POEMS, Amyloidosis, ongoing plasma cell leukemia (PCL)
3. History of Human Immunodeficiency Virus (HIV)
4. Active, uncontrolled HBV infection despite antiviral therapy.
5. Uncontrolled cardiac, pulmonary, gastrointestinal (GI), hepatic, renal, central nervous system(CNS) diseases not due to myeloma, at the discretion of investigator, that are not a candidate for T cell engager (TCE) therapy
6. Uncontrolled or recurrent infections
7. Autoimmune disease requiring systemic treatment (except for low dose steroids, equivalent to 10mg/day or less of prednisone)
8. Disabling psychiatric conditions, substance abuse (alcohol, or drug), dementia, altered mental status
9. Any other active malignancies within 5 years of completing treatment (with the exception of hormonal therapies for breast or prostate cancer) and >minimal risk of recurrence
10. Myelodysplastic syndromes (MDS)
11. Any issues that may impair the ability of the participant to receive or tolerate the planned treatment, to understand the informed consent, or any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant or that would prevent, limit, or confound the protocol specified assessments.
12. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Elra or other agents used in study.
13. History or possible non-compliance with recommended treatments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-07-14 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Christine Ye, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org